CLINICAL TRIAL: NCT04951817
Title: Using 68Ga-PSMA PET/CT for the Assessment of Osseous Tumor Burden in mCRPC Patients Undergoing 223Ra-dichloride Injections
Brief Title: 68Ga-PSMA PET/CT for Ra223 Assessment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jing-Ren Tseng, MD, PhD, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202002133A0
Record Dates: First submitted 2021-06-30; First posted 2021-07-07 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Prostate Cancer
Keywords: Prostate Cancer; Treatment response; Ra223; Ga-68 PSMA Ligand; Bone scan
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ga68-PSMA ligand (Experimental): Glass vial with 5~20 mCi(185-740 MBq) of 68Ga-PSMA ligand in ≤10% EtOH with aqueous sterile water for injection solution (approximately 15.5 mL), ≧ 0.33 mCi/mL @ EOS。
  Interventions: Drug: Ga-68 PSMA ligand

INTERVENTIONS:
Drug: Ga-68 PSMA ligand — For PET/CT PSMA scan, the subject will have catheter(s) placed for intravenous administration of [68Ga]PSMA-11. Subjects will receive a single intravenous bolus of 2-5 mCi [68Ga]PSMA-11 and received PET/CT scan 60 minutes later.PSMA PET-CT scan was performed on a GE Discovery MI PET/CT system.
  Other Names: Ga68-PSMA-11 (Gallium-68 labeled HBED-CC PSMA)

SUMMARY:
Primary objective:

i.The primary objective is to compare the diagnostic positivity in progression of 68Ga-PSMA PET and Bone scan.

Secondary objectives:

i.The correlation between PET osseous tumor burden index and Alk-P level ii.The correlation between PET osseous tumor burden index and PSA level

DETAILED DESCRIPTION:
It is a open-label single-arm clinical trial. Outcome measurement is the positivity rate of Ga68-PSMA-11 PET-defined progression and Bone Scan-defined progression. The primary objective is to compare the diagnostic positivity in progression of PSMA PET and BS. The 2×2 contingency table with four diagnostic outcomes (both positive, PET positive/BS negative, PET negative/BS positive, and both negative) will be conducted based on the enrolled subjects. Both diagnostic tools (Ga68-PSMA-11 PET and BS) are applied to a given set of individuals. Since both diagnostic tools will performed on each subject, then paired data result and methods that account for the correlated binary outcomes are necessary. McNemar's test will be used to compare the positivity of the two tools. Assuming that Ga68-PSMA-11 PET in patients detect more metastatic lesions/progression by 26.5% (i.e. p10-p01=0.265) and the discordant percentage is 38.5 % (i.e. p10+p01=0.385). Under the hypothesis H0: p10=p01, achieving an 80% power at the 5% of significance level, the sample size is 44. Based on expecting 15% of missing rate, the adjusted sample size will be 52. This calculation was done by PASS software (Power Analysis and Sample Size version 11.0.8, NCSS, Kaysville, Utah, USA).

For PET/CT PSMA scan, the subject will have catheter(s) placed for intravenous administration of [68Ga]PSMA-11. Subjects will receive a single intravenous bolus of 2-5 mCi [68Ga]PSMA-11 and received PET/CT scan 60 minutes later. PSMA PET-CT scan was performed on a GE Discovery MI PET/CT system. The CT scan parameters were 120 kVp, 30 mA to 300 mA acquired with auto mA , 40× 0.625 collimator configuration, and pitch of 0.984 : 1. All images were reconstructed with a 500 mm field of view and a slice thickness of 5 mm. The PET acquisition time was 3 mins per bed position with maximum overlap (35 slices). Images were reconstructed using Q clear with beta value of 550, PSF correction, and non-TOF (QCHD-S). The matrix is 256 × 256. After image acquisition, the subject will be observed for half an hour, and will be discharged if no adverse event happens. EKG, blood and biochemistry test will be performed before and after first PET scan no more than two weeks. Except baseline Ga68-PSMA-11 PET/CT scan, patients will receive serial PET scans after 3rd injection of Ra-233 and 6th injection of Ra-223. All of the images were interpreted by an experienced nuclear medicine physicians.

ELIGIBILITY:
Inclusion Criteria:

1. Males with 40-85 years of age and life expectancy more than 3 months
2. Patient was diagnosed as mCRPC, and meet the standard criteria of using 223Ra-dichloride (symptomatic bone metastasis, at least two bone metastasis sites, no visceral organ metastasis)
3. Willing to sign the informed consent
4. ECOG performance status Grade 0-2

Exclusion Criteria:

1. Unable to tolerate the PET/CT scan, such as those with claustrophobia, unable to lie still, consciousness unclear, vital sign unstable.
2. With renal impairment (glomerular filtration rate lower than 30 ml/min/1.73 m2), and allergy to medium contrast.
3. Significant abnormal lab data (AST or ALT more than three times of normal value), and high risk to conduct examination after evaluations of PI.
4. Patient had previous other malignancy history
5. Patient experiences grade 3-4 neutropenia (neutrophil counts less than 1000/uL) or thrombocytopenia (platelet counts less than 50x103/uL) lasting > 14 days

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patient only
Enrollment: 52 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change of lesion detection number by PET imaging | 9-11 weeks or 21-23 weeks
  Lesion detection number before and under Ra223 therapy on the PSMA PET imaging with a time interval 9-11 weeks and/or 21-23 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Ren Tseng, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital ,Linkou, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No